CLINICAL TRIAL: NCT00140699
Title: Balance Control and Maturation in Normal and Deaf Children Aged From 6 to 14 Years Old
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Other Study IDs: 2001.264
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Deaf Children
Keywords: Children, Hearing loss, Balance control, Sensory inputs
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Balance

SUMMARY:
Balance disorders in children are poorly known, underestimated, and rarely assessed. Technologies to assess balance in children are almost non-existent, apart from a few exceptions. Such technologies are routinely used in adults for some decades, and are of considerable contribution in the diagnosis and treatment of adults balance disorders.

The aim of this study is :

1. to assess objectively children balance disorders.
2. to provide technologies suitable for children balance assessement.
3. to study children balance disorders suffering from sensorineural hearing loss.

DETAILED DESCRIPTION:
The inner ear included two sensorineural organs closely linked: the cochlea and the vestibule. With regards to children inner ear affliction, only cochlear function is taken into consideration, whereas balance related to vestibule function is often neglected.

Congenital sensorineural hearing loss is frequent (3/1000 births, Martin et al. 1981, Fortum et al. 1997). Furthermore, otitis media is among the most frequent afflictions discovered in small childhood, and Handicaps secondary to sensorineural hearing loss are numerous: language, cognitive disorders, delay according to school and social integration (Joint Commitee on Infant Hearing 1994, Casselbrant et al. 2005, Jung et al. 2005).

In counterpart, children balance disorders are often unknown and underestimated. However, they clinically lead to an evident handicap in case of acute or chronic otitis media (Caselbrant et al. 1995). Balance control involves three sensory systems tightly linked: vision, vestibule, and somesthesia. From the links between vision and vestibule originate the visio-vestibular and vestibulo-ocular reflexes (VVOR,VOR). Dynamic Posturography (DP) is a technology able to measure each of these sensory inputs involved in balance control by recording sensory organization test (SOT). This technology is available for adults for a few decades but are poorly used in children (Wiener-Vacher et al. 1996, 1998, Casselbrant et al 1995, 2005).

Aims:

1-To assess objectively children balance control (to provide normative data according to the age). 2- to put in place methods to investigate children balance disorders. 3- to study children balance disorders suffering from sensorineural hearing loss.

Methods:

Studied population: two groups of children are involved and compared in this study: 150 healthy children and 150 children suffering from sensorineural hearing loss. Each group is divided into three age groups: 6-8, 8-10, 10-12 years old.

Assessment:

The following parameters are recorded in both groups: VVOR and VOR, SOT on two DP Equitest and Balance Quest. Transient Evoked Otoacoustic Emissions were recorded too in order to prove normal hearing status in the healthy group and hearing loss in the sensorineural hearing loss group.

ELIGIBILITY:
Inclusion Criteria:

Healthy group :

* Normal neurological status
* Normal visual status
* Normal ENT status
* TEOE present
* Informed consent aproved and signed

Sensorineural hearing loss group :

* Normal neurological status
* Normal visual status
* Otitis media or endocochlear hearing loss
* In the case of otitis, flat curve at tympanometry
* Transmissional aspect at BAERs
* Informed consent aproved and signed

Ages: 6 Years to 14 Years | Sex: All
Age Groups: Child
Enrollment: 240

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Ferber-Viart, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France